CLINICAL TRIAL: NCT02784327
Title: A Single-Dose, Open-Label, Multi-Center Study to Evaluate the Safety, Pharmacokinetics and Preliminary Efficacy of PRF110 in Bunionectomy Surgery
Brief Title: A Study to Evaluate the Safety, Pharmacokinetics and Preliminary Efficacy of PRF110 in Bunionectomy Surgery
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: PainReform LTD (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRF110-102
Record Dates: First submitted 2016-05-24; First posted 2016-05-27 (Estimated); Last update posted 2016-05-27 (Estimated); Status verified 2016-05

CONDITIONS: Post Operative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- PRF110- oily solution (Experimental): Post-operative application of new extended release PRF110- oily solution (Ropivacaine)
  Interventions: Drug: PRF110

INTERVENTIONS:
Drug: PRF110
  Other Names: Ropivacaine oily solution

SUMMARY:
PRF110 is new extended release oily solution formulation of ropivacaine that is intended for local infiltration into surgical wounds. The purpose of this study is to determine the safety and early efficacy of PRF110 in bunionectomy surgery, to measure the pharmacokinetic profile of PRF110 over 72 hours and evaluate the duration of analgesia witnessed in the surgical setting.

DETAILED DESCRIPTION:
PRF110 is new extended release oily solution formulation of ropivacaine that is intended for local infiltration into surgical wounds. The formulation is designed to slowly release the ropivacaine over 36-72 hours. By providing local analgesia over a long time span, the need for systemic analgesics is expected to be reduced. The purpose of this study is to determine the safety and early efficacy of PRF110 in bunionectomy surgery, to measure the pharmacokinetic profile of PRF110 over 72 hours and evaluate the duration of analgesia witnessed in the surgical setting.

ELIGIBILITY:
Inclusion Criteria:

1. Able to provide written informed consent prior to any study procedures;
2. Able to communicate clearly with the Investigators and study staff;
3. Males and females aged between 18 - 85 years of age;
4. Scheduled for elective primary unilateral first metatarsal bunionectomy surgery (osteotomy and internal fixation) with no collateral procedures;
5. Females must be physically incapable of childbearing potential (postmenopausal for more than at least 2 years or surgically sterile) or practicing an acceptable method of contraception (hormonal, barrier with spermicide, intrauterine device, vasectomized partner, or abstinence). Subjects using hormonal birth control must have received at least 1 cycle of treatment prior to study drug administration. At Baseline, all females of childbearing potential must have a negative pregnancy test and not be breast feeding;
6. Negative urine drug screen for drugs of abuse at Screening and on Day 1 prior to surgery; a positive drug screen result may be permitted if the subject has been on a stable dose of an allowed medication for >30 days (antipsychotics, antiepileptics, sedatives, hypnotics, antianxiety agents, or antidepressants);
7. American Society of Anesthesiologists (ASA) risk class of I to II;
8. Body Mass Index ≤32.

Exclusion Criteria:

1. Has known allergies to an opioid, unless has subsequently tolerated other opioids and, in the opinion of the Investigator, could tolerate a rescue drug containing fentanyl;
2. Has a known or suspected allergy to paracetamol, ibuprofen or dipyrone;
3. Has a known or suspected allergy to any local anesthetic;
4. Has atrial fibrillation/flutter, an inserted pacemaker, or complete left bundle branch block (LBBB) on ECG; or myocardial infarction within 6 months prior to surgery;
5. Has a clinically significant abnormal ECG at screening;
6. Has a known or suspected history of diagnosed alcohol, opiate or other substance abuse within 12 months prior to screening;
7. Is unable to refrain from alcohol consumption for a period beginning 24 hours prior to surgery through the end of the 72 hour evaluation period;
8. Has taken any analgesic within 12 hours or any aspirin-containing product within 7 days of the Baseline assessments;
9. Has taken any opioid analgesics or used systemic steroids within 4 days of surgery;
10. Has been using opiates or any non-steroidal anti-inflammatory drug chronically (more than 10 consecutive days) anytime over the past 3 months;
11. Has used antipsychotics, antiepileptics, sedatives, hypnotics, antianxiety agents or antidepressants for < 30 days prior to surgery or had a dose change within the previous 30 days;
12. Has taken any prescription or over-the-counter medication within 4 days prior to surgery that, in the opinion of the Investigator, could potentially confound the analgesic response;
13. Has taken herbal agents or nutraceuticals during any of the 7 days prior to surgery that, in the opinion of the Investigator, could potentially confound the analgesic response;
14. Has any clinically significant condition or a significant laboratory abnormality that would, in the opinion of the Investigator, preclude study participation;
15. Unable or unwilling, in the opinion of the Investigator to comply with the requirements of the protocol;
16. Has received another investigational drug within 30 days of scheduled surgery;
17. Has donated blood within three months prior to start of the study;
18. Employees of the Investigator and study site or the sponsor, as well as family members of the employees or the investigator or the sponsor.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2016-08; Primary Completion 2017-04 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment emergent adverse events | 10 days
  All adverse events (AE) reported by the subjects will be recorded throughout the trial period

SECONDARY OUTCOMES:
Time to first rescue medication | 72 hours
  Time to first rescue medication
Total amount of rescue medication used during the study | 10 days
  Total amount of rescue medication used during the study
Pain intensity recorded at rest | 72 hours
  Pain intensity which will be recorded at rest at Hours 1, 2, 4, 6, 8, 10, 12, 18 (optional) 24, 28, 32, 36, 48, 52, 56, 60 and 72.
Subject global assessment of PRF110 | 72 hours
  Subject global assessment which will be recorded at Hours 24, 48 and 72.

OTHER OUTCOMES:
PRF110 plasma concentrations | 72 hours
  Samples will be collected at designated times up to 72hrs post drug application

CONTACTS AND LOCATIONS:
Overall Officials: Shai Efrati, Dr., Principal Investigator — Assaf-Harofeh Medical Center; Natan Bruck, Dr., Principal Investigator — The Chaim Sheba Medical Center
Locations (2):
- Israel (2):
  - The Chaim Sheba Medical Center, Ramat Gan
  - Assaf Harofeh Medical Center, Ẕerifin